CLINICAL TRIAL: NCT07367438
Title: Effect of Subthreshold Stimulation on Fatigability, Lower Limb Muscle Function and Strength, and Inflammatory Blood Markers in Patients With Rheumatoid Arthritis: A Randomized Controlled Study.
Brief Title: Effect of Subthreshold Stimulation on Fatigue in Rheumatoid Arthritis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Ayman Mohamed, PhD, MSc, DPT, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BNS3
Record Dates: First submitted 2026-01-18; First posted 2026-01-26 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: Subthreshold stimulation; Fatigability; lower limb strength; Inflammatory Blood Markers
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): This group will receive subthreshold stimulation
  Interventions: Device: Subthreshold stimulation
- Control group (Sham Comparator): This group will not receive any treatment
  Interventions: Other: Sham treatment

INTERVENTIONS:
Device: Subthreshold stimulation — The study group received subthreshold stimulation via a two-channel portable electrical stimulation unit (BTL-4620, Czech Republic). Two self-adhesive electrodes (9 × 5 cm Axelgaard PALS, Axelgaard Manufacturing Co. Ltd., CA, USA) were used to deliver a premixed amplitude-modulated electrical current with 100 Hz frequency/pulse 60ms width. Four electrodes were placed on the quadriceps muscle to include all the muscle as follows: the first electrode was placed on proximal third, the the secod electrode was placed on middle third, the third electrode was placed on distal lateral third, and the fourth electrode was placed on the distal medial third. Before applying the electrodes, the skin of the anterior thigh was cleansed with alcohol to decrease the surface impedance. The intensity of the device gradually increased till the participant started to feel the electrical current. Then, the intensity was decreased by 10%. Therefore, the intensity is about 90% of the sensation threshold.
  Arms: Study group
Other: Sham treatment — The device will be placed on the patient without any stimulation
  Arms: Control group

SUMMARY:
The study will include 2 groups. The study group will receive subthreshold stimulation, while the control group will receive sham treatment.

DETAILED DESCRIPTION:
This study will investigate the effect of subthreshold stimulation on fatigue-related parameters in patients with rheumatoid arthritis. This study will include 2 groups Study and the control group. The outcome measures will include Fatigability, Lower Limb Muscle Function and Strength, and Inflammatory Blood Markers. The measurements will be performed at the baseline, after 8 weeks, and after 12 weeks (follow-up).

ELIGIBILITY:
Inclusion Criteria:

* Sixty patients with rheumatoid arthritis based on physician diagnosis and referral.

  * The patients' ages ranged from 30 to 55 (Tedeschi et al., 2013).
  * Body mass index ranged from 25-30 kg/m2.
  * Patients diagnosed with rheumatoid arthritis 5 years ago.

Exclusion Criteria:

* Patients had chronic heart failure, cancer, chronic kidney disease, infection, and any other autoimmune disease (García-Morales et al., 2020).

  * Patients had unstable ischemic heart disease or arrhythmia (Lange et al., 2019).
  * Patients had joint surgery within 6 months before inclusion which did not allow them to perform physical activity as arthroplasty (Lange et al., 2019).
  * Patients had received biologics for RA treatments (Lange et al., 2019).

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Fatigability | 8 weeks
  Lower limb muscle performance was measured using an isokinetic dynamometer (Biodex Medical INC., Shirley, New York, USA). It was used to assess peak torque, total work, average power, work fatigue percentage, and agonist-antagonist ratio. This instrument is a gold standard, valid, objective, and reliable system used in research, clinical testing, and rehabilitation
C-reactive protein blood | 8 weeks
  C-reactive protein blood test is a gold standard, reliable, and valid adequate operation technique (Spasovski and Sotirova, 2014). C-reactive protein is an inexpensive and readily available biomarker to assess systemic inflammation and clinical outcomes in RA. C-reactive protein is measured from a blood sample that comes from a vein. The result is expressed in milligrams per liter (mg/L). The report might indicate that the level is high, low, or normal. Most healthy adults have CRP levels lower than 0.3 mg/L. Clinical trials often specify elevated CRP for ≥6 mg/L (

SECONDARY OUTCOMES:
Functional disability | 8 weeks
  The investigatorswill use the Health Assessment Questionnaire to measures functional disability through patient self-reports across eight categories (dressing, arising, eating, walking, hygiene, reach, grip, activities) using a 0-3 scale (no difficulty to unable to do)
Rheumatoid Arthritis Pain | 8 weeks
  The Rheumatoid Arthritis Pain Scale (RAPS) is a validated, 24-item, self-report questionnaire designed to capture the multidimensional pain experience in rheumatoid arthritis (RA) patients, assessing physiological, affective (emotional), sensory-discriminative, and cognitive aspects of pain through a single score, helping clinicians understand pain beyond just intensity for better treatment planning. Developed from pain theories, RAPS uses Likert scales, with items scored 0 (never) to 6 (always) for a total score range of 0-144, offering a comprehensive tool for assessing pain's impact and treatment effectiveness.

IPD SHARING:
Plan to Share IPD: Undecided